CLINICAL TRIAL: NCT03939936
Title: Effects of Non-surgical Periodontal Therapy on Inflammatory Markers of Psoriasis
Brief Title: The Effect of Periodontal Treatment on Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozge Gokturk (Other)
Responsible Party: Sponsor-Investigator, Ozge Gokturk, Principal Investigator, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17-KAEK-44
Record Dates: First submitted 2019-04-26; First posted 2019-05-07 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Periodontal Diseases
Keywords: Psoriasis
MeSH Terms: conditions — Periodontal Diseases; Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Active Comparator): Psoriatic measurements and saliva samples were taken from periodontal disease patients before treatment and after 8 weeks.
  Intervention: Non-surgical periodontal treatment was performed and the Psoriasis Area and Severity Index (PASI) was filled, saliva samples were taken.
  Interventions: Other: Psoriatic measurements; Other: Non-surgical periodontal treatment; Other: saliva samples
- Control Group (Placebo Comparator): Psoriatic measurements and saliva samples were taken from periodontal disease patients at the baseline and after 8 weeks without the periodontal treatment.
  Intervention: Psoriasis Area and Severity Index (PASI) was filled, saliva samples were taken.
  Interventions: Other: Psoriatic measurements; Other: saliva samples

INTERVENTIONS:
Other: Psoriatic measurements — Psoriasis Area and Severity Index (PASI) was performed baseline and after 8 weeks. Saliva samples were taken from patients for the evaluation of proinflammatory cytokine baseline and after 8 weeks.
Other: Non-surgical periodontal treatment — Non-surgical periodontal treatment was performed baseline and after 8 weeks. Saliva samples were taken from patients for the evaluation of proinflammatory cytokine baseline and after 8 weeks.
  Arms: Test Group
Other: saliva samples — Saliva samples were taken from patients for the evaluation of proinflammatory cytokine baseline and after 8 weeks.

SUMMARY:
There is a relationship between psoriasis and periodontal disease. This relationship may be double-sided.

DETAILED DESCRIPTION:
The aim of this randomized controlled clinical study was to determine the effect of non-surgical mechanical periodontal treatment on psoriasis. The study population consisted of 92 periodontitis patients with psoriasis who had untreated periodontal disease. Two randomized groups were formed from these patients. Immediate periodontal treatment (test group, n = 46) and delayed periodontal treatment (control group, n = 46). Clinical periodontal measures, saliva interleukin 2, interleukin 6 and secretory immunoglobulin A levels and PASI scores were performed at baseline and 8th week in control and test group.

ELIGIBILITY:
Inclusion Criteria:

* the presence at least 20 remaining teeth,
* the presence of Stage I or Stage II Periodontitis,
* the presence of diagnosed psoriasis.

Exclusion Criteria:

* patients who had the immune-inflammatory disease and require antibiotic prophylaxis,
* patients who received periodontal treatment prior to 6 months,
* women who were breastfeeding or pregnant,
* patients using medicines such as antibiotics, anti-inflammatory drugs, immune-suppressants.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Proinflammatory cytokines | Baseline and after 8 weeks
  The changes in proinflammatory cytokines levels within 8 weeks. Higher values represent a worse outcome. The decrease in proinflammatory cytokines levels is expected after periodontal treatment.

SECONDARY OUTCOMES:
Gingival index | Baseline and after 8 weeks
  The changes in gingival index level after periodontal treatment. Gingival index was measured for determining the severity of disease and clinical outcome. Higher values represent a worse outcome. After periodontal treatment, a reduction in gingival index value is expected.
PASI index | Baseline and after 8 weeks
  The changes in PASI index level after periodontal treatment. PASI index was measured for determining the severity of psoriasis disease. Higher values represent a worse outcome. After periodontal treatment, a reduction in PASI index value is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Atiye Ogrum, Principal Investigator — Gaziosmanpasa Universty
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No